CLINICAL TRIAL: NCT02342730
Title: Referral of Obese Endometrial Cancer Survivors to a Bariatric Specialist and a Healthier Survivorship: A Prospective Intervention Cohort Study
Brief Title: Weight Loss Referral for Healthier Survivorship in Obese Stage I-II Endometrial Cancer Survivors or Atypical Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE13813; NCI-2014-02477 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE13813 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Complex Endometrial Hyperplasia With Atypia; Stage IA Uterine Corpus Cancer; Stage IB Uterine Corpus Cancer; Stage II Uterine Corpus Cancer
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight Loss Referral (Experimental): Patients are referred to a weight loss specialist for assistance with weight loss and medical chart reviews are performed at baseline and every 3 months for 24 months. Patients complete Quality-of-Life Assessment (EORTC- QLQ-C30 and EORTC-QLQ-EN24) at baseline, 12, and 24 months. Patients are also contacted at 90 days to determine whether they have initiated any weight loss interventions.
  Interventions: Behavioral: Weight Loss Specialist; Other: Quality-of-Life Assessment; Other: Medical Chart Review

INTERVENTIONS:
Behavioral: Weight Loss Specialist — Referred to a weight loss specialist
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Intervention
Other: Quality-of-Life Assessment — Complete EORTC-QLQ questionnaires
  Other Names: Quality of Life Assessment
Other: Medical Chart Review — Chart reviews are performed
  Other Names: Chart Review

SUMMARY:
This pilot clinical trial studies whether obese stage I-II endometrial cancer survivors or patients with atypical hyperplasia (abnormal cells in the lining of the uterus) would go see a weight loss specialist if it was recommended by their cancer doctor. Excess body weight or obesity is one of the most common contributors to (causes of) endometrial cancer. Over two-thirds of women who have survived endometrial cancer are obese. Complications of obesity, such as heart disease are often more dangerous than the cancer itself. A weight loss of even 5-10% of excess body weight is associated with improved health. Often, meeting with a doctor or person who is an expert in weight loss (bariatric specialist) is the best way to lose weight and keep it off. Endometrial cancer survivors or patients with atypical hyperplasia who go see a weight loss specialist recommended by their doctor may be able to achieve a healthier body weight.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I.Our primary outcome for the purposes of the pilot study will be to describe recruitment in terms of accrual (number of subjects who agree to participate) and compliance (number of patients who follow up with the obesity referral). This will be described in terms of a specific number as well as a rate.

* Accrual rate is the number of women accrued divided by the number of women approached for the study.
* Compliance rate is the number of women who comply with the referral divided by the number of women accrued.

Several secondary outcomes will be described:

* Weight loss at 12 & 24 months.
* Obesity interventions implemented (medical, surgical, behavioral, and selfguided)
* The incidence of obesity related comorbidities at baseline and 12 and 24 months (myocardial infarction, venous thromboembolism, stroke, diabetes and hypertension.)
* Cancer specific outcomes (recurrence rate, progression free survival).
* Mortality otucomes (Overall survival, cause of death)
* In patients with diabetes, we will record the number of diabetic medications required and the most recent hemoglobin A1C.
* In patients with hypertension, we will record the number of antihypertensive medications required
* We will assess the level of functioning, quality of life and symptomatology of women at baseline, 12 and 24 months using the EORTC-QLQ-C30 and EORTC-QLQ-EN24.

  * Primary and secondary outcomes will be compared in relation to the timing of the referral by the gynecologic oncologist (within 1 year or greater than 1 year out from the endometrial cancer/hyperplasia diagnosis).
  * Secondary outcomes of subjects included in this study will be compared to a historic cohort matches for age, stage and BMI in a 2:1 fashion.

OUTLINE:

Patients are referred to a weight loss specialist for assistance with weight loss and chart reviews are performed at baseline and every 3 months for 24 months. Patients complete the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire (QLQ)-Cancer (C)30 and EORTC-QLQ-Endometrial Cancer (EN)24 at baseline, 12, and 24 months. Patients are also contacted at 90 days to determine whether they have initiated any weight loss interventions.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of stage I or II endometrial cancer or a diagnosis of complex atypical hyperplasia
* BMI of at least 30 kg/msq

Exclusion Criteria:

* Advanced disease (stage III or greater)
* Recurrent or progressive endometrial cancer
* Non endometrioid histology (such as serous uterine cancer or uterine carcinosarcoma)
* History of bariatric surgery for weight loss
* Ongoing medically supervised weight loss (under the care of a physician)
* Poorly controlled psychiatric or medical conditions
* Active second primary malignancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-12-17; Primary Completion 2015-05-18 (Actual); Study Completion 2015-05-18 (Actual)

PRIMARY OUTCOMES:
Accrual with intervention, defined as number of subjects who agree to participate | Up to 24 months
  Descriptive statistics will be used. Will be compared using chi square or fisher exact tests.
Compliance with intervention, defined as number of patients who follow up with the obesity referral | Up to 24 months
  Descriptive statistics will be used. Will be compared using chi square or fisher exact tests.

SECONDARY OUTCOMES:
Weight loss (in kilograms) | Baseline to 12 months
  Descriptive statistics will be used. Will compare groups using a paired t-test.
Weight loss (in kilograms) | Baseline to 24 months
  Descriptive statistics will be used. Will compare groups using a paired t-test.
Compliance with lifestyle changes (based on affirmative response to 3 month follow up when asked if lifestyle changes have been adopted) | At 3 months
  Will be compared using chi square or fisher exact tests.
Incidence of obesity related comorbidities and adverse events (diabetes, hypertension, myocardial infarction, stroke, venous thromboembolism) | Baseline
  Descriptive statistics will be used to detail incidence of new major health events (myocardial infarction, stroke, new diabetes diagnosis, new venous thromboembolism, new hypertension diagnosis, death, date of death, cause of death). The occurrence new major health events and cancer related events will be compared using chi square or fisher exact tests.
Incidence of obesity related comorbidities and adverse events (diabetes, hypertension, myocardial infarction, stroke, venous thromboembolism) | At 12 months
  Descriptive statistics will be used to detail incidence of new major health events (myocardial infarction, stroke, new diabetes diagnosis, new venous thromboembolism, new hypertension diagnosis, death, date of death, cause of death). The occurrence new major health events and cancer related events will be compared using chi square or fisher exact tests.
Incidence of obesity related comorbidities and adverse events (diabetes, hypertension, myocardial infarction, stroke, venous thromboembolism) | At 24 months
  Descriptive statistics will be used to detail incidence of new major health events (myocardial infarction, stroke, new diabetes diagnosis, new venous thromboembolism, new hypertension diagnosis, death, date of death, cause of death). The occurrence new major health events and cancer related events will be compared using chi square or fisher exact tests.
Progression free survival | Up to 24 months
  Descriptive statistics will be used. Will be described with Kaplan Meier curves.
Overall survival | Up to 24 months
  Descriptive statistics will be used. Will be described with Kaplan Meier curves.
Recurrence rate | Up to 24 months
  Descriptive statistics will be used to detail cancer related outcomes (cancer recurrence, date and location of recurrence, cancer related death).
Level of functioning, quality of life, and symptomatology, as measured by the EORTC-QLQ-C30 and EORTC-QLQ-EN24 | At 12 months
  Will compare groups using a paired t-test.
Level of functioning, quality of life, and symptomatology, as measured by the EORTC-QLQ-C30 and EORTC-QLQ-EN24 | At 24 months
  Will compare groups using a paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Jernigan, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States